CLINICAL TRIAL: NCT06485115
Title: The Effectiveness of Combining a Home-based Digital Motor Telerehabilitation Program With Conventional Therapy in Progressive Multiple Sclerosis: a Multicentre, Randomized Controlled Trial
Brief Title: Telerehabilitation in Progressive Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Marialuisa Gandolfi, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/R-Multi/010
Record Dates: First submitted 2024-06-17; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Balance; Dual Task; Cognitive Function; Digital Telemedicine; Wearables
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Digital motor Telerehabilitation added to conventional therapy (Experimental): All patients will receive an individualized ten sessions of an in-hospital rehabilitation program (1 hour/day, 3 days/week) by a qualified physiotherapist at each participating unit. Then, the EG will follow a 12-week individualized Digital Telerehabilitation program (1 hour/day, 3 days/week, EG).
  Interventions: Device: Digital Telerehabilitation (Euleria Home); Other: Conventional therapy
- Conventional therapy alone (Other): All patients will receive an individualized ten sessions of an in-hospital rehabilitation program (1 hour/day, 3 days/week) by a qualified physiotherapist at each participating unit. Then, the CG will not receive any additional therapy except for general instructions for self- management according to the allocation group.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: Digital Telerehabilitation (Euleria Home) — After the in-hospital rehabilitation treatment (1 h/day, 3 days/week), the EG patients will perform the Digital Telerehabilitation program at home. The three weekly sessions will be asynchronous (with the caregiver's supervision if necessary). At each Unit, the physiotherapist will develop the training sessions on the Home- based Digital Telerehabilitation program and monitor the training execution provided by the digital device to adapt the rehabilitation treatment to the patients' improvements/difficulties. The Digital Telerehabilitation device (Euleria Home, Euleria Health) will consist of one wearable sensor and an app on a tablet that guides the patient through the customized exercise-therapy path configured by the professional. The sensor is worn on different body segments to monitor movements and provides real-time feedback on angles, balance, and repetitions.
  Arms: Home-based Digital motor Telerehabilitation added to conventional therapy
Other: Conventional therapy — After the in-hospital rehabilitation treatment (1 h/day, 3 days/week), the CG patients will be advised to perform the Self-management activities learned during the in-hospital rehabilitation training without home-based Digital Telerehabilitation devices.

SUMMARY:
Multiple sclerosis (MS) is a highly disabling chronic, inflammatory, demyelinating disease of the Central Nervous System (CNS). Significant progress has been made during the past three decades in managing the relapsing-remitting phase of Multiple Sclerosis (RRMS). However, once patients have entered the progressive stage of MS (secondary progressive, SPMS), therapeutic options are limited to symptomatic treatments and rehabilitation. In addition, 10-20% of patients experience unremitting disease progression (primary progressive MS, or PPMS). The limited research focusing on Progressive MS (PMS) and the lack of ecological validity highlight the need for a bolder approach that combines more than one intervention intending to produce synergistic effects. The primary aim is to test the effectiveness of combining a home-based Digital Telerehabilitation program with in-hospital rehabilitation on mobility against in-hospital rehabilitation alone.

DETAILED DESCRIPTION:
The literature emphasizes a striking dearth of studies devoted solely to people with SPMS or PPMS and the lack of ecological validity in assessing the results. This suggests that an additional effort is required, a bolder approach that combines more than one intervention intending to produce synergistic effects, an improvement in one area boosting the putative benefits of therapy in another, the overall outcome exceeding the sum of the individual treatments.

The primary aim will be to test the effectiveness of combining a home-based digital motor telerehabilitation program (experimental intervention) with in-hospital rehabilitation on mobility (primary outcome) against in-hospital rehabilitation without any additional therapy except for general instructions for self-management as usual care (conventional treatment) in patients with SPMS or PPMS.

The secondary aims will be to explore the effects on measures of motor and cognitive function; the patients reported outcomes on balance and upper extremity function, fatigue, pain, anxiety, and depressive symptoms; the self-perception of clinical change; and Health-Related Quality of Life. Furthermore, the investigators will explore the patient's perspective and experience with Digital Telerehabilitation post-treatment using quantitative-qualitative methods (EG intervention). An economic evaluation of the introduction of the digital telemedicine program will be carried out within the health technology assessment (HTA) framework, considering the perspective of the healthcare system and society as a whole.

This single-blind RCT with 2-parallel arms will compare the effects between the experimental group (EG) and control group (CG). After the screening, an administrator external to research groups (the principal investigator) will generate a block randomization list at each Unit to prevent selection bias using an automated randomization system (www.randomization.com) (allocation ratio 1:1) to assign eligible patients to either the EG or the CG. Patients will be stratified according to the EDSS (≥ 6 and < 6). Group allocation will be kept concealed. All patients will receive an individualized ten sessions of an in-hospital rehabilitation program (1 hour/day, 3 days/week) by a qualified physiotherapist at each participating unit. Then, the EG will follow a 12-week individualized Digital Telerehabilitation program (1 hour/day, 3 days/week, EG) while the CG will not receive any additional therapy except for general instructions for self-management according to the allocation group. All the patients will undergo four clinical evaluations: before (T0) and after (T1) the in-hospital rehabilitation program, 12 weeks (T2), and 24 weeks (follow-up, T3) after it. One researcher assistant with experience in assessing primary and secondary outcomes blinded to group assignment will evaluate study participants at all time points in each Unit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75;
* Diagnosis of MS (primary or secondary progressive);
* Mild to moderate balance impairments with increased fall risk, defined as TUG > 8.4s;
* A disability rate, as calculated using the Kurtzke Expanded Disability Status Scale (EDSS) lower than 7;
* Acceptable level of digital skills;
* The presence of the caregiver.

Exclusion Criteria:

* Other conditions that may affect motor function;
* Impaired cognitive functioning (Mini-Mental Status Examination <24/30);
* Severe visual deficits (daltonism and visual acuity deficit);
* Unable or refused to attend the rehabilitation treatment.

Patients who fulfill the following specified inclusion criteria will also undergo an EEG evaluation. However, ineligibility for this examination does not exclude them from participating in the rehabilitation study.

The inclusion criteria for the EEG protocol will include:

* The absence of metallic implants in the brain;
* No history of brain surgery;
* No use of medications that alter cortical excitability or are presumed to affect brain plasticity;
* Right-handed dominance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Timed Up and Go test | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The patient mobility will be measured by the Timed Up and Go (TUG) test (Euleria Lab, Rovereto - TN, Italy). We will give patients verbal instructions to stand up from a chair, walk 3 meters, cross a line marked on the floor, turn around, walk back, and sit down.

SECONDARY OUTCOMES:
Change in the Multiple Sclerosis Functional Composite (MSFC) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Multiple Sclerosis Functional Composite (MSFC) is a multidimensional, three-component performance scale to assess the degree of impairment in MS patients: gait, upper extremity function, and cognition. Since the units of three variables measured by three tests are different (Timed 25-foot Walk Test (T25FW) and 9-Hole Peg Test (9HPT) and number of correct answers in 3-second version of the Paced Auditory Serial Addition Test (PASAT-3)), raw scores should be converted to a common metric, namely z-scores. The overall composite score (MSFC score) is calculated by adding the z-scores for each test. Component scores are entered into a formula with scores from the reference population in order to derive the means and standard deviations required to determine Z-scores. A score of +1 indicates that, on average, an individual scored 1 SD better than the reference population and a score of -1 indicates that an individual scored 1 SD worse than the reference population.
Mental workload through Electroencephalography (EEG) during Multiple Sclerosis Functional Composite Score | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  During the Multiple Sclerosis Functional Composite (MSFC) administration, the participant's brain activity will be recorded using electroencephalography (EEG) to assess the participant's mental workload and vigilance state during the task.
Vigilance state through Electroencephalography (EEG) during Multiple Sclerosis Functional Composite Score | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  During the Multiple Sclerosis Functional Composite (MSFC) administration, the participant's brain activity will be recorded using electroencephalography (EEG) to assess the participant's vigilance state during the task.
Surface electromyography (EMG) during the performance of the Nine Hole Peg test part of the Multiple Sclerosis Functional Composite (MSFC). | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The muscular activity of the upper limb will be recorded using surface electromyography (EMG) system during the performance of the Nine Hole Peg test part of the Multiple Sclerosis Functional Composite (MSFC).
Inertial Measurement Unit (IMU) system during the performance of the Nine Hole Peg test part of the Multiple Sclerosis Functional Composite (MSFC). | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The kinematics of the upper limb will be recorded using Inertial Measurement Unit (IMU) system during the performance of the Nine Hole Peg test part of the Multiple Sclerosis Functional Composite (MSFC).
Change in the Fatigue Severity Scale (FSS) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Fatigue Severity Scale (FSS) is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations. The items are scored on a 7 point scale (1= strongly disagree and 7= strongly agree). The minimum score is 9 and maximum score possible is 63. Higher score indicate greater fatigue severity.
Change in the Activities-specific balance confidence (ABC) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Activities-specific balance confidence (ABC) Scale is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. It is a 16-item self-report measure in which patients rate their balance confidence for performing activities. Items are rated on a rating scale that ranges from 0 - 100. Score of zero represents no confidence, a score of 100 represents complete confidence. Overall score is calculated by adding item scores and then dividing by the total number of items.
Change in the Manual Ability Measure-36 (MAM-36) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Manual Ability Measure-36 (MAM-36) is designed as an outcome instrument to assess hand function based on the patient's responses to functional questions. Patient rates functional abilities based on his or her perception of the difficulty or ease in completing one or two-handed daily tasks. Item level scores are as follows: 1=cannot do, 2=very hard, 3=a little hard and 4=easy, 0=not applicable/almost never do. The total score ranging from 0 to 144; higher scores indicate better-perceived manual ability.
The number of falls in the previous month | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Number of falls in the previous month
Timed Up and Go (TUG) test - Cognitive | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  In the Timed Up and Go (TUG) test - Cognitive, individuals will be asked to complete the test while counting backward by threes from a randomly selected number between 20 and 100
Electroencephalography (EEG) during the Timed Up and Go (TUG) test - Cognitive | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  During the Timed Up and Go (TUG) test - Cognitive, the participant's brain activity will be recorded using electroencephalography (EEG) to assess the participant's mental workload and vigilance state during the task
Timed Up and Go (TUG) test - Manual | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  In the Timed Up and Go (TUG) test - Manual, individuals will be asked to complete the test holding a cup filled with water.
Electroencephalography (EEG) during the Timed Up and Go (TUG) test - Manual | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  During the Timed Up and Go (TUG) test - Manual, the participant's brain activity will be recorded using electroencephalography (EEG) to assess the participant's mental workload and vigilance state during the task
Change in the gait speed (cm/s) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Gait analysis will be used to collect gait speed (cm/s)
Change in the cadence (step/min) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Gait analysis will be used to collect cadence (step/min)
Change in the stride length (cm) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Gait analysis will be used to collect stride length (cm)
Change in the length of the centre of pressure (CoP) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Stabilometric platform will be used to evaluated the length of the centre of pressure (CoP)
Change in the trajectory (mm) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Stabilometric platform will be used to evaluated the trajectory (mm)
Change in the sway area (mm2) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Stabilometric platform will be used to evaluated the sway area (mm2)
Change in the Brief Pain Inventory (BPI) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Brief Pain Inventory (BPI) is a self-administered questionnaire divided into intensity (range: 0-40; higher = worse) and interference (range: 0-70; higher = worse)
Change in the Hospital Anxiety and Depression Scale | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Hospital Anxiety and Depression Scale (HADS) is a brief self-report questionnaire composed of 14 items (7 items each for anxiety and depression), with a score ranging between 0 and 21 for the anxiety and depression subscales. Scores between 8 and 10 indicate a moderate presence of symptoms, whereas a score greater than 11 indicates a significant number of symptoms that likely correspond with a clinical diagnosis.
Change in the Hospital Anxiety and Depression Scale - Anxiety (HADS-A) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Hospital Anxiety and Depression Scale - Anxiety (HADS-A, 7 items) subscale scores will be calculated, possibly ranging from 0 (no symptoms) to 21 (most severe symptoms)
Change in the Hospital Anxiety and Depression Scale - Depression (HADS-D) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Hospital Anxiety and Depression Scale - Depression (HADS-D, 7 items) subscale scores will be calculated, possibly ranging from 0 (no symptoms) to 21 (most severe symptoms)
Change in the Modified Asworth Scale | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Modified Ashworth Scale is a 6-points muscle tone assessment scale used to assess the resistance experienced during passive range of motion. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity.
Change in the Modified Tardieu Scale | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Modified Tardieu Scale si a clinical measure of muscle spasticity in patients with neurological conditions. The Modified Tardieu Scale comprises four elements, including R1, R2, R2-R1 and X score. R1 represents an angle of catch, where a sudden increase of muscle resistance is felt during a fast passive stretch. R2 is an angle indicating the tested muscle length at a slow passive range of motion. R2-R1 was introduced to differentiate spasticity from contracture.15 Contracture is indicated if the value of R2-R1 is small, while a large value indicates spasticity. The X score describes types of muscle resistance when passive stretches are applied during the assessment (grade 0-5). Quality of Muscle Reaction (scored 0-5); 0 is no resistance to passive ROM to 5 indicating joint is immobile.
Change in the the Multiple Sclerosis Quality Of Life-54 (MSQOL-54) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The summary scores are the physical health composite summary and the mental health composite summary. The single item measures are satisfaction with sexual function and change in health. There is no single overall score for the MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores.
The EuroQol five domains (EQ-5D) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The EuroQol five-dimensions (EQ5D) is a versatile quality of life (QOL) instrument with five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a visual analog scale. It can be used to calculate quality-adjusted life years. The scale ranges from 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state' or 'the worst health you can imagine').
The volumes of health services | Before treatment (T0), and 24 weeks after the in-hospital treatment (T3)
  The volumes of health services will be collected at baseline encompassing the resources use 6 months prior the start of the study and 24 weeks after the in-hospital treatment (T3) estimating the resource use during the entire trial duration
The Multiple Sclerosis Health Resource Utilization Survey (MS-HRS) | Before treatment (T0), and 24 weeks after the in-hospital treatment (T3)
  Direct healthcare costs will be assessed using the Multiple Sclerosis Health Resource Utilization Survey (MS-HRS). The Multiple Sclerosis Health Resource Utilization Survey (MS-HRS) is a multilingual, reliable, valid and easy to administer questionnaire providing a holistic cross-sectional and longitudinal assessment of resource utilization in people with multiple sclerosis.
The TheiTA Productivity Cost Questionnaire | Before treatment (T0), and 24 weeks after the in-hospital treatment (T3)
  Indirect costs will be measured using validated log as the TheiTA Productivity Cost Questionnaire for productivity loss
Change in the Clinical Global Impression (CGI) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Self-rated perception of change will be assessed with the 7-point Clinical Global Impression (CGI) scale with scores from 1 (very much improved) to 7 (very much worse)
Changes in effective brain connectivity through Electroencephalography (EEG) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  Only patients eligible for EEG will be evaluated to detect changes in effective brain connectivity through EEG during a motor observation, execution, and motor imagery task.
Change in the Brief Illness Perception Questionnaire (B-IPQ) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Brief Illness Perception Questionnaire (B-IPQ) consists of eight items on an individual's cognitive and emotional representation of one's health conditions.To score the B-IPQ questionnaire, each item is rated on a 0-10 scale, with higher scores indicating a more threatening perception of the illness. The total score is calculated by summing the scores of all eight items, with a possible range of 0-80. Higher scores indicate worse illness perception.
Change in the Multidimensional Psychological Flexibility Inventory (MPFI) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Multidimensional Psychological Flexibility Inventory (MPFI), a 60-item scale that measures the 6 dimensions of psychological flexibility and the 6 dimensions of inflexibility posited by the Hexaflex model. To score the Multidimensional Psychological Flexibility Inventory subscales, are assigned responses point values from 1 to 6 and then average the responses across the items of each scale so that higher scores reflect higher levels of the dimension being assessed by each set of items. The averages of the 6 flexibility subscales can be averaged to create a composite representing global flexibility. Similarly, the averages of the 6 inflexibility subscales can be averaged to create a global inflexibility composite.
Change in the Self-Efficacy for Multiple Sclerosis Scale (SEMS) | Before treatment (T0), after 4 weeks of in-hospital rehabilitation (T1), at the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2), and 24 weeks after the in-hospital treatment (T3)
  The Self-Efficacy for Multiple Sclerosis Scale (SEMS) assesses self-efficacy related to the management of MS. It comprises 15 items starting from the root statement "I am confident that I can…" and is rated on a 5-point Likert scale from 0 (Not at all confident) to 4 (Very confident)
Tele-healthcare Satisfaction Questionnaire-Wearable Technology | At the end of the 12 weeks of telerehabilitation
  Tele-healthcare Satisfaction Questionnaire-Wearable Technology consists of 6 areas (benefit, usability, self-concept, privacy and loss of control, quality of life, and wearing comfort) that evaluate the satisfaction of the subject with the wearable part of a system. Each area includes 5 statements rated by the user on a 5-point Likert scale between 0 (strongly disagree with the statement) and 4 (strongly agree with the statement)
Patients' In-home Digital Telerehabilitation training experience questionnaire | At the end of the 12 weeks of telerehabilitation
  One questionnaire used by the research group to evaluate patients' In-home Digital Telerehabilitation training experience with the Digital Telerehabilitation program "EG treatment experience". The questionnaire consists of 9 questions scored on a 10-point scale (1=not at all; 10=very much) and 17 open-ended questions to investigate pleasantness, usefulness, acceptability, safety, satisfaction, and future development.
Activity levels through Technology-based Objective Measures (TOMS) | After 4 weeks of in-hospital rehabilitation (T1), At the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2)
  Wearable sensors (Axivity AX3) will be used to collect the activity levels.
Number of steps through Technology-based Objective Measures (TOMS) | After 4 weeks of in-hospital rehabilitation (T1), At the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2)
  Wearable sensors (Axivity AX3) will be used to collect the number of steps.
Distance traveled through Technology-based Objective Measures (TOMS) | After 4 weeks of in-hospital rehabilitation (T1), At the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2)
  Wearable sensors (Axivity AX3) will be used to collect the distance traveled.
Risk of fall assessment | During the 4 weeks in-hospital rehabilitation (3 days/week for 4 week - total of 10 sessions)
  An inertial sensor will be used to detect near falls during balance training and i twill be placed on the forehead with an elastic band.
Adverse Events | At the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2)
  Safety in terms of reported adverse events during the treatment (falls or event near falling) will be collected
Number of patients who accept/refuse the treatment | At the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2)
  Measures of feasibility in terms of the recruitment rate before the end of treatment will be collected.
Number of dropouts | At the end of the 12 weeks of telerehabilitation or usual care after the end of the in-hospital treatment (T2)
  Measures of feasibility in terms of the number of dropouts before the end of treatment will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Marialuisa Gandolfi, Principal Investigator — Universita di Verona
Locations (1):
- Department of Neurosciences, Biomedicine and Movement Sciences, University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lassmann H, Bruck W, Lucchinetti CF. The immunopathology of multiple sclerosis: an overview. Brain Pathol. 2007 Apr;17(2):210-8. doi: 10.1111/j.1750-3639.2007.00064.x. PMID 17388952
- [Background] Lublin FD, Reingold SC. Defining the clinical course of multiple sclerosis: results of an international survey. National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. Neurology. 1996 Apr;46(4):907-11. doi: 10.1212/wnl.46.4.907. PMID 8780061
- [Background] Lassmann H, van Horssen J, Mahad D. Progressive multiple sclerosis: pathology and pathogenesis. Nat Rev Neurol. 2012 Nov 5;8(11):647-56. doi: 10.1038/nrneurol.2012.168. Epub 2012 Sep 25. PMID 23007702
- [Background] Feinstein A, Freeman J, Lo AC. Treatment of progressive multiple sclerosis: what works, what does not, and what is needed. Lancet Neurol. 2015 Feb;14(2):194-207. doi: 10.1016/S1474-4422(14)70231-5. PMID 25772898
- [Background] Morgen K, Kadom N, Sawaki L, Tessitore A, Ohayon J, McFarland H, Frank J, Martin R, Cohen LG. Training-dependent plasticity in patients with multiple sclerosis. Brain. 2004 Nov;127(Pt 11):2506-17. doi: 10.1093/brain/awh266. Epub 2004 Sep 29. PMID 15456705
- [Background] Tomassini V, Matthews PM, Thompson AJ, Fuglo D, Geurts JJ, Johansen-Berg H, Jones DK, Rocca MA, Wise RG, Barkhof F, Palace J. Neuroplasticity and functional recovery in multiple sclerosis. Nat Rev Neurol. 2012 Nov 5;8(11):635-46. doi: 10.1038/nrneurol.2012.179. PMID 22986429
- [Background] Tieri G, Morone G, Paolucci S, Iosa M. Virtual reality in cognitive and motor rehabilitation: facts, fiction and fallacies. Expert Rev Med Devices. 2018 Feb;15(2):107-117. doi: 10.1080/17434440.2018.1425613. Epub 2018 Jan 10. PMID 29313388
- [Background] Peran P, Nemmi F, Dutilleul C, Finamore L, Falletta Caravasso C, Troisi E, Iosa M, Sabatini U, Grazia Grasso M. Neuroplasticity and brain reorganization associated with positive outcomes of multidisciplinary rehabilitation in progressive multiple sclerosis: A fMRI study. Mult Scler Relat Disord. 2020 Jul;42:102127. doi: 10.1016/j.msard.2020.102127. Epub 2020 May 6. PMID 32438326
- [Background] Lotze M, Ladda AM, Stephan KM. Cerebral plasticity as the basis for upper limb recovery following brain damage. Neurosci Biobehav Rev. 2019 Apr;99:49-58. doi: 10.1016/j.neubiorev.2019.01.027. Epub 2019 Jan 30. PMID 30710580
- [Background] Schmidt R, Lee T, Winstein C, et al. Motor control and learning: a behavioral emphasis. 2018. cited Sep. 17, 2022.,36
- [Background] Gandolfi M, Mazzoleni S, Morone G, Iosa M, Galletti F, Smania N. The role of feedback in the robotic-assisted upper limb rehabilitation in people with multiple sclerosis: a systematic review. Expert Rev Med Devices. 2023 Jan;20(1):35-44. doi: 10.1080/17434440.2023.2169129. Epub 2023 Jan 29. PMID 36649574
- [Background] Dehem S, Montedoro V, Edwards MG, Detrembleur C, Stoquart G, Renders A, Heins S, Bruno D, Lejeune T. Development of a robotic upper limb assessment to configure a serious game. NeuroRehabilitation. 2019;44(2):263-274. doi: 10.3233/NRE-182525. PMID 31006692
- [Background] Maier M, Rubio Ballester B, Duff A, Duarte Oller E, Verschure PFMJ. Effect of Specific Over Nonspecific VR-Based Rehabilitation on Poststroke Motor Recovery: A Systematic Meta-analysis. Neurorehabil Neural Repair. 2019 Feb;33(2):112-129. doi: 10.1177/1545968318820169. Epub 2019 Jan 30. PMID 30700224
- [Background] Shaw MT, Best P, Frontario A, Charvet LE. Telerehabilitation benefits patients with multiple sclerosis in an urban setting. J Telemed Telecare. 2021 Jan;27(1):39-45. doi: 10.1177/1357633X19861830. Epub 2019 Jul 15. PMID 31307269
- [Background] Thompson AJ. Neurorehabilitation in multiple sclerosis: foundations, facts and fiction. Curr Opin Neurol. 2005 Jun;18(3):267-71. doi: 10.1097/01.wco.0000169743.37159.a0. PMID 15891410
- [Background] Freeman J, Hendrie W, Jarrett L, Hawton A, Barton A, Dennett R, Jones B, Zajicek J, Creanor S. Assessment of a home-based standing frame programme in people with progressive multiple sclerosis (SUMS): a pragmatic, multi-centre, randomised, controlled trial and cost-effectiveness analysis. Lancet Neurol. 2019 Aug;18(8):736-747. doi: 10.1016/S1474-4422(19)30190-5. PMID 31301748
- [Background] Gandolfi M, Munari D, Geroin C, Gajofatto A, Benedetti MD, Midiri A, Carla F, Picelli A, Waldner A, Smania N. Sensory integration balance training in patients with multiple sclerosis: A randomized, controlled trial. Mult Scler. 2015 Oct;21(11):1453-62. doi: 10.1177/1352458514562438. Epub 2015 Jan 12. PMID 25583852
- [Background] Straudi S, Tramontano M, Russo EF, et al. Robot-assisted upper limb training for patients with multiple sclerosis: an evidence-based review of clinical applications and effectiveness. Appl Sci. 2021 Dec;12(1):2222.
- [Background] Munari D, Fonte C, Varalta V, Battistuzzi E, Cassini S, Montagnoli AP, Gandolfi M, Modenese A, Filippetti M, Smania N, Picelli A. Effects of robot-assisted gait training combined with virtual reality on motor and cognitive functions in patients with multiple sclerosis: A pilot, single-blind, randomized controlled trial. Restor Neurol Neurosci. 2020;38(2):151-164. doi: 10.3233/RNN-190974. PMID 32333564
- [Background] Gandolfi M, Vale N, Dimitrova EK, Mazzoleni S, Battini E, Benedetti MD, Gajofatto A, Ferraro F, Castelli M, Camin M, Filippetti M, De Paoli C, Chemello E, Picelli A, Corradi J, Waldner A, Saltuari L, Smania N. Effects of High-intensity Robot-assisted Hand Training on Upper Limb Recovery and Muscle Activity in Individuals With Multiple Sclerosis: A Randomized, Controlled, Single-Blinded Trial. Front Neurol. 2018 Oct 24;9:905. doi: 10.3389/fneur.2018.00905. eCollection 2018. PMID 30405526
- [Background] Vale N, Gandolfi M, Mazzoleni S, Battini E, Dimitrova EK, Gajofatto A, Ferraro F, Castelli M, Camin M, Filippetti M, De Paoli C, Picelli A, Corradi J, Chemello E, Waldner A, Saltuari L, Smania N. Characterization of Upper Limb Impairments at Body Function, Activity, and Participation in Persons With Multiple Sclerosis by Behavioral and EMG Assessment: A Cross-Sectional Study. Front Neurol. 2020 Feb 14;10:1395. doi: 10.3389/fneur.2019.01395. eCollection 2019. PMID 32116983
- [Background] Gandolfi M, Geroin C, Picelli A, Munari D, Waldner A, Tamburin S, Marchioretto F, Smania N. Robot-assisted vs. sensory integration training in treating gait and balance dysfunctions in patients with multiple sclerosis: a randomized controlled trial. Front Hum Neurosci. 2014 May 22;8:318. doi: 10.3389/fnhum.2014.00318. eCollection 2014. PMID 24904361
- [Background] Baroni A, Fregna G, Milani G, Severini G, Zani G, Basaglia N, Straudi S. Video game therapy on mobility and dual tasking in multiple sclerosis: study protocol for a randomised controlled trial. BMJ Open. 2021 Oct 21;11(10):e052005. doi: 10.1136/bmjopen-2021-052005. PMID 34675018
- [Background] Straudi S, De Marco G, Martinuzzi C, Baroni A, Lamberti N, Brondi L, Da Roit M, Pizzongolo LDM, Basaglia N, Manfredini F. Combining a supervised and home-based task-oriented circuit training improves walking endurance in patients with multiple sclerosis. The MS_TOCT randomized-controlled trial. Mult Scler Relat Disord. 2022 Apr;60:103721. doi: 10.1016/j.msard.2022.103721. Epub 2022 Mar 5. PMID 35276451
- [Background] Kalron A, Dolev M, Givon U. Further construct validity of the Timed Up-and-Go Test as a measure of ambulation in multiple sclerosis patients. Eur J Phys Rehabil Med. 2017 Dec;53(6):841-847. doi: 10.23736/S1973-9087.17.04599-3. Epub 2017 Mar 13. PMID 28290192
- [Background] Fischer JS, Rudick RA, Cutter GR, Reingold SC. The Multiple Sclerosis Functional Composite Measure (MSFC): an integrated approach to MS clinical outcome assessment. National MS Society Clinical Outcomes Assessment Task Force. Mult Scler. 1999 Aug;5(4):244-50. doi: 10.1177/135245859900500409. PMID 10467383
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Solaro C, Di Giovanni R, Grange E, Brichetto G, Mueller M, Tacchino A, Bertoni R, Patti F, Pappalardo A, Prosperini L, Castelli L, Rosato R, Cattaneo D, Marengo D. Italian translation and psychometric validation of the Manual Ability Measure-36 (MAM-36) and its correlation with an objective measure of upper limb function in patients with multiple sclerosis. Neurol Sci. 2020 Jun;41(6):1539-1546. doi: 10.1007/s10072-020-04263-2. Epub 2020 Jan 23. PMID 31974795
- [Background] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Background] Guy W. (1976). Clinical global impression scale. The ECDEU Assessment Manual for Psychopharmacology, Revised. US Department of Health, Education, and Welfare Publication (ADM), 76(338), 218-222. Rockville, MD: National Institute of Mental Health
- [Background] Buchholz I, Janssen MF, Kohlmann T, Feng YS. A Systematic Review of Studies Comparing the Measurement Properties of the Three-Level and Five-Level Versions of the EQ-5D. Pharmacoeconomics. 2018 Jun;36(6):645-661. doi: 10.1007/s40273-018-0642-5. PMID 29572719
- [Background] Donisi V, Gajofatto A, Mazzi MA, Gobbin F, Busch IM, Ghellere A, Klonova A, Rudi D, Vitali F, Schena F, Del Piccolo L, Rimondini M. A Bio-Psycho-Social Co-created Intervention for Young Adults With Multiple Sclerosis (ESPRIMO): Rationale and Study Protocol for a Feasibility Study. Front Psychol. 2021 Feb 23;12:598726. doi: 10.3389/fpsyg.2021.598726. eCollection 2021. PMID 33708157
- [Background] Donisi V, Poli S, Mazzi MA, Gobbin F, Schena F, Del Piccolo L, Bigardi V, Gajofatto A, Rimondini M. Promoting participatory research in chronicity: The ESPRIMO biopsychosocial intervention for young adults with multiple sclerosis. Front Psychol. 2022 Nov 3;13:1042234. doi: 10.3389/fpsyg.2022.1042234. eCollection 2022. PMID 36405126
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Rolffs JL, Rogge RD, Wilson KG. Disentangling Components of Flexibility via the Hexaflex Model: Development and Validation of the Multidimensional Psychological Flexibility Inventory (MPFI). Assessment. 2018 Jun;25(4):458-482. doi: 10.1177/1073191116645905. Epub 2016 May 5. PMID 27152011
- [Background] Bonino, S., Graziano, F., Borghi, M., Marengo, D., Molinengo, G., Calandri, E. (2018). The self-efficacy in Multiple Sclerosis (SEMS) Scale: development and validation with Rasch analysis. European Journal of Psychological Assessment, 34 (5), 352-360. DOI: 10.1027/1015-5759/a000350
- [Background] Emilia Ambrosini, Simona Ferrante, Mauro Rossini, Franco Molteni, Margit Gföhler, Werner Reichenfelser, Alexander Duschau-Wicke, Giancarlo Ferrigno and Alessandra Pedrocchi (2014). Functional and usability assessment of a robotic exoskeleton arm to support activities of daily life. Robotica, 32, pp 1213-1224 Doi:10.1017/S0263574714001891.
- [Background] Carpinella I, Cattaneo D, Bonora G, Bowman T, Martina L, Montesano A, Ferrarin M. Wearable Sensor-Based Biofeedback Training for Balance and Gait in Parkinson Disease: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Apr;98(4):622-630.e3. doi: 10.1016/j.apmr.2016.11.003. Epub 2016 Dec 10. PMID 27965005
- [Background] Kim YK, Park E, Lee A, Im CH, Kim YH. Changes in network connectivity during motor imagery and execution. PLoS One. 2018 Jan 11;13(1):e0190715. doi: 10.1371/journal.pone.0190715. eCollection 2018. PMID 29324886
- [Background] Ness NH, Haase R, Kern R, Schriefer D, Ettle B, Cornelissen C, Akguen K, Ziemssen T. The Multiple Sclerosis Health Resource Utilization Survey (MS-HRS): Development and Validation Study. J Med Internet Res. 2020 Mar 17;22(3):e17921. doi: 10.2196/17921. PMID 32181745
- [Background] Marques E, Johnson EC, Gooberman-Hill R, Blom AW, Noble S. Using resource use logs to reduce the amount of missing data in economic evaluations alongside trials. Value Health. 2013 Jan-Feb;16(1):195-201. doi: 10.1016/j.jval.2012.09.008. PMID 23337231
- [Background] www.imta.nl iMTA Productivity and Health Research Group. Manual iMTA Medical Cost Questionnaire (iMCQ). Rotterdam: iMTA, Erasmus University Rotterdam, 2018
- [Background] Bouwmans C, Krol M, Severens H, Koopmanschap M, Brouwer W, Hakkaart-van Roijen L. The iMTA Productivity Cost Questionnaire: A Standardized Instrument for Measuring and Valuing Health-Related Productivity Losses. Value Health. 2015 Sep;18(6):753-8. doi: 10.1016/j.jval.2015.05.009. Epub 2015 Aug 20. PMID 26409601
- [Background] Sciaraffa N, Di Flumeri G, Germano D, Giorgi A, Di Florio A, Borghini G, Vozzi A, Ronca V, Babiloni F, Arico P. Evaluation of a New Lightweight EEG Technology for Translational Applications of Passive Brain-Computer Interfaces. Front Hum Neurosci. 2022 Jul 14;16:901387. doi: 10.3389/fnhum.2022.901387. eCollection 2022. PMID 35911603
- [Background] Wiendl H, Hohlfeld R. Multiple sclerosis therapeutics: unexpected outcomes clouding undisputed successes. Neurology. 2009 Mar 17;72(11):1008-15. doi: 10.1212/01.wnl.0000344417.42972.54. PMID 19289741